CLINICAL TRIAL: NCT01059786
Title: Randomized Phase II Trial of Rituximab With Either Pentostatin or Bendamustine for Multiply Relapsed or Refractory Hairy Cell Leukemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Robert Kreitman, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 100025; 10-C-0025
Record Dates: First submitted 2010-01-29; First posted 2010-02-01 (Estimated); Results first posted 2024-05-01 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Hairy Cell Leukemia
Keywords: Monoclonal Antibody; Purine Analog; Soluble CD25; Minimal Residual Disease MRD; CD20
MeSH Terms: conditions — Leukemia, Hairy Cell; Neoplasm, Residual | interventions — Pentostatin; Rituximab; Bendamustine Hydrochloride; Acetaminophen; Diphenhydramine; Epinephrine; Histamine Antagonists; Adrenal Cortex Hormones; Bronchodilator Agents; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Arm 1 - Non-Randomized to 70 mg/m^2 Bendamustine-Rituximab (Experimental): Rituximab + Bendamustine at 70 mg/m^2 for initial tolerability study (closed)
  Interventions: Drug: Rituximab; Drug: Bendamustine; Drug: Acetaminophen; Drug: Diphenhydramine; Drug: Epinephrine; Drug: Antihistamines; Drug: Corticosteroids; Drug: Bronchodilators; Other: Intravenous (IV) Saline
- Arm 2 - Non-randomized to 90 mg/m^2 Bendamustine-Rituximab (Experimental): Rituximab + Bendamustine at 90 mg/m^2 for initial tolerability study (closed)
  Interventions: Drug: Rituximab; Drug: Bendamustine; Drug: Acetaminophen; Drug: Diphenhydramine; Drug: Epinephrine; Drug: Antihistamines; Drug: Corticosteroids; Drug: Bronchodilators; Other: Intravenous (IV) Saline
- Arm 3 - Randomized to 90 mg/m^2 Bendamustine-Rituximab (Active Comparator): Rituximab + Bendamustine (at the tolerated dose)
  Interventions: Drug: Rituximab; Drug: Bendamustine; Drug: Acetaminophen; Drug: Diphenhydramine; Drug: Epinephrine; Drug: Antihistamines; Drug: Corticosteroids; Drug: Bronchodilators; Other: Intravenous (IV) Saline
- Arm 4 - Randomized to Pentostatin-Rituximab (Active Comparator): Rituximab + Pentostatin
  Interventions: Drug: Pentostatin; Drug: Rituximab; Drug: Acetaminophen; Drug: Diphenhydramine; Drug: Epinephrine; Drug: Antihistamines; Drug: Corticosteroids; Drug: Bronchodilators; Other: Intravenous (IV) Saline
- Non-randomized to Bendamustine 90mg/m^2 or Pentostatin 4mg/m^2 with Rituximab (Experimental): After initial tolerability studies are completed. Non-randomize up to 4 total participants to Bendamustine and/or Pentostatin with Rituximab
  Interventions: Drug: Pentostatin; Drug: Rituximab; Drug: Bendamustine; Drug: Acetaminophen; Drug: Diphenhydramine; Drug: Epinephrine; Drug: Antihistamines; Drug: Corticosteroids; Drug: Bronchodilators; Other: Intravenous (IV) Saline

INTERVENTIONS:
Drug: Pentostatin — 28 participants to pentostatin 4 mg/m^2 days 1 and 15 of each cycle.
  Other Names: Nipent
  Arms: Arm 4 - Randomized to Pentostatin-Rituximab; Non-randomized to Bendamustine 90mg/m^2 or Pentostatin 4mg/m^2 with Rituximab
Drug: Rituximab — Rituximab 375 mg/m^2 on day 1, 15 for 6 x 28-day cycles
  Other Names: Rituxan
Drug: Bendamustine — 1-4 participants to bendamustine 90 mg/m^2/day, days 1 and 2 each cycle
  Other Names: Bendeka; Treanda
  Arms: Arm 1 - Non-Randomized to 70 mg/m^2 Bendamustine-Rituximab; Arm 2 - Non-randomized to 90 mg/m^2 Bendamustine-Rituximab; Arm 3 - Randomized to 90 mg/m^2 Bendamustine-Rituximab; Non-randomized to Bendamustine 90mg/m^2 or Pentostatin 4mg/m^2 with Rituximab
Drug: Acetaminophen — Treatment of infusion-related symptoms with acetaminophen is recommended.
  Other Names: Tylenol
Drug: Diphenhydramine — Treatment of infusion-related symptoms with diphenhydramine is recommended.
  Other Names: Benadryl
Drug: Epinephrine — Epinephrine should be available for immediate use in the event of a hypersensitivity reaction to Rituximab.
  Other Names: Adrenaline
Drug: Antihistamines — Antihistamines should be available for immediate use in the event of a hypersensitivity reaction to Rituximab.
Drug: Corticosteroids — Corticosteroids should be available for immediate use in the event of a hypersensitivity reaction to Rituximab.
  Other Names: Corticoid
Drug: Bronchodilators — Additional treatment with bronchodilators may be indicated.
  Other Names: Broncholytic
Other: Intravenous (IV) Saline — Additional treatment with intravenous (IV) saline may be indicated.

SUMMARY:
Background:

* Researchers are attempting to develop new treatments for hairy cell leukemia (HCL) that has not responded well to or has recurred after standard HCL therapies. One nonstandard treatment for HCL is rituximab, an antibody that binds to the cancer cells and helps the immune system destroy them. By combining rituximab with other anti-cancer drugs, researchers hope to determine whether the combined drugs are successful in treating HCL.
* Pentostatin and bendamustine are two anti-cancer drugs that have been used to treat different kinds of blood and immune system cancers. Bendamustine is approved to treat other kinds of leukemia and lymphoma, but it has not been used to treat HCL. Pentostatin has been used for more than 20 years to treat HCL, but it has not been combined with rituximab in official clinical trials.

Objectives:

* To determine whether rituximab with either pentostatin or bendamustine is a more effective treatment for HCL than rituximab alone.
* To determine whether pentostatin or bendamustine is a more effective treatment for HCL when combined with rituximab.

Eligibility:

- Individuals at least 18 years of age who have been diagnosed with hairy cell leukemia that has not responded well to or has relapsed after standard HCL therapies.

Design:

* The study will last for four treatment cycles of 28 days each.
* Prior to the study, participants will be screened with a full medical history and physical exam, bone marrow biopsy (if one has not been performed in the last 6 months), computed tomography (CT) or ultrasound scan, tumor measurements, and other tests as required by the researchers. Participants will provide blood and urine samples at this time as well.
* Rituximab with bendamustine: Participants will receive rituximab on Days 1 and 15 of each cycle and bendamustine on Days 1 and 2 of each cycle, for a total of four cycles.
* Rituximab with pentostatin: Participants will receive rituximab on Days 1 and 15 of each cycle and pentostatin on rituximab on Days 1 and 15 of each cycle, for a total of four cycles.
* Participants will have regular tests during the treatment cycles, including bone marrow biopsies and CT or ultrasound scans. Participants will also provide regular blood and urine samples to assess the results of treatment.

DETAILED DESCRIPTION:
Background:

* Hairy cell leukemia (HCL) is highly responsive to purine analogs cladribine and pentostatin, without evidence of cure. Neither is standard after 2 courses, due to cumulative marrow and T-cell toxicity and declining remission rates and durations. Once resistant, patients after multiple relapses can die of disease-related cytopenias.
* Rituximab alone in 51 patients from 5 trials who had cytopenias and at least 1 prior purine analog resulted in 10 complete + 10 partial remissions (complete response (CR) + partial response (PR) = overall response rate (ORR 39%).
* Rituximab with cladribine gives high CR rates in 1st or 2nd line but is not standard.
* While cladribine use is more common for 1st and 2nd line, pentostatin is often used for subsequent treatment because of < 100% cross-resistance.
* Retrospective published data for pentostatin plus rituximab in HCL include 7 of 7 responses with 6 (86%) CRs, and there are no prospective data.
* Recombinant immunotoxins targeting cluster of Differentiation 25 (CD25) (LMB-2) and cluster of differentiation-22 (CD22) (CAT-3888 (BL22) and R490A (HA22) are highly active in purine analog resistant HCL. Palliative pentostatin-rituximab is often used off-protocol for patients with immunogenicity needing more therapy.
* Bendamustine is approved for early treatment of chronic lymphocytic leukemia (CLL) and is effective with rituximab for relapsed/refractory CLL. Its use in HCL is unreported.
* CRs with minimal residual disease (MRD) by immunohistochemistry (IHC) of bone marrow biopsy (BMBx IHC), can relapse early. Tests for HCL MRD in blood or marrow include flow cytometry (fluorescence-activated cell sorting (FACS) or polymerase chain reaction (PCR) using consensus primers. The most sensitive MRD test in HCL is real-time quantitative PCR using sequence-specific primers (real-time quantitative polymerase chain reaction (RQ-PCR).
* Of 5 HCL-specific trials listed on Cancer.gov, 2 are phase II trials of cladribine + rituximab in 1st and 2nd line (1 randomized at National Institutes of Health (NIH), 1 non-randomized at MDA), and 3 NIH phase I-II trials of recombinant immunotoxins BL22, HA22 and LMB-2.

Objectives:

-Primary:

--To determine if pentostatin + rituximab and bendamustine + rituximab are each associated with adequate response rates (ORR=PR+CR) in patients with relapsed HCL, and, if so, to select which combination is likely to be superior.

Eligibility:

* HCL needing therapy, either greater than or equal to 2 prior courses of purine analog, 1 course purine analog plus greater than or equal to 1 course rituximab if < 1 year response to the 1 course purine analog, diagnosis of HCL variant (HCLv), or unmutated immunoglobulin heavy variable 4-34 (IGHV4-34+) expressing HCL/HCLv.
* Prior treatment, ineligibility for, or patient refusal of recombinant immunotoxin.

Design:

* Rituximab 375 mg/m^2 on day 1, 15 for 6 x 28-day cycles (all 72 patients).
* Initial tolerability study: 12 patients receive rituximab + bendamustine (nonrandom), including 6 at 70 mg/m^2 and 6 at 90 mg/m^2 of bendamustine.
* Randomize: 1) 28 patients to bendamustine 90 mg/m^2/day, days 1 and 2 each cycle 2) 28 patients to pentostatin 4 mg/m^2 days 1 and 15 of each cycle.
* Non-randomized: up to 4 patients to receive either bendamustine 90 mg/m^2P2P/day, days 1 and 2 each cycle or pentostatin 4 mg/m^2P2P days 1 and 15 of each cycle.
* Statistics: If > 14/28 respond, can conclude with 90% power that response > 40% in that arm. >80% probability of selecting the better arm if true response probability is approximately 40-50% on the inferior arm and >15% higher on the superior arm.
* Stratify to equalize the % of patients/arm refractory to last course of purine analog.
* Accrual Ceiling: 72 evaluable participants

ELIGIBILITY:
* INCLUSION CRITERIA:
* Evidence of Hairy Cell Leukemia (HCL) by flow cytometry of blood or a solid (lymph node) mass, confirmed by the Laboratory of Pathology, National Cancer Institute (NCI), including positivity for cluster of Differentiation 19 (CD19), cluster of differentiation-22 (CD22), cluster of differentiate 20 (CD20), and Integrin, alpha X (CD11c). Patients with flow cytometry consistent with hairy cell leukemia-variant (HCLv) are eligible, including those with cluster of Differentiation 25 (CD25) and/or cluster of differentiation 103 (CD103) negative disease.
* bone marrow biopsy (BMBx) or bone marrow aspiration (BMA) consistent with HCL, confirmed by National Institutes of Health (NIH) Laboratory of Pathology, NCI, or the Department of Laboratory Medicine, Clinical Center, NIH, unless the diagnosis can be confirmed from a solid (lymph node) mass.
* Treatment indicated based on demonstration of at least one of the following, no more than 4 weeks from the time of enrollment, and no less than 6 months after prior cladribine and no less than 4 weeks after other prior treatment, if applicable.

  * Neutropenia (Absolute neutrophil count (ANC) less than 1000 cells/microl).
  * Anemia (Hemoglobin (Hgb) less than 10g/dL).
  * Thrombocytopenia (Platelet (PLT) less than 100,000/microl).
  * Absolute lymphocyte count (ALC) of greater than 5,000 cells/microL
  * Symptomatic splenomegaly.
  * Enlarging lymph nodes greater than 2cm.
  * Repeated infections requiring oral or intravenous (i.v.) antibiotics.
  * Increasing lytic bone lesions

Patients who have eligible blood counts within 4 weeks from enrollment will not be considered ineligible if subsequent blood counts prior to enrollment fluctuate and become ineligible up until the time of enrollment.

* One of the following:

  * At least 2 prior courses of purine analog
  * 1 prior course of purine analog plus greater than or equal to1 course of rituximab if the response to the course of purine analog lasted less than 1 year.
  * Diagnosis of HCL variant (HCLv)
  * Unmutated (>98% homology to germline) immunoglobulin heavy variable 4-34 (IGHV4-34+) expressing hairy cell leukemia (HCL)/HCLv
* Eastern Cooperative Oncology Group (ECOG) performance status (102) of 0-3
* Patients must be able to understand and give informed consent.
* Creatinine less than or equal to 1.5 or creatinine clearance greater than or equal to 60 ml/min.
* Bilirubin less than or equal to 2 unless consistent with Gilbert's (total/direct greater than 5), alanine transaminase (ALT) and aspartate aminotransferase (AST) less than or equal to 3 x upper limits of normal.
* No other therapy (i.e., chemotherapy, interferon) for 4 weeks prior to study entry, or cladribine for 6 months prior to study entry, unless progressive disease more than 2 months after cladribine is documented.
* Age at least 18
* Men and women of reproductive potential must agree to use an acceptable method of birth control during treatment and for twelve months after completion of treatment.
* Patients must be willing to co-enroll in the investigators companion protocol 10-C-0066 titled Collection of Human Samples to Study Hairy Cell and other Leukemias, and to Develop Recombinant Immunotoxins for Cancer Treatment.

EXCLUSION CRITERIA:

* Presence of active untreated infection
* Uncontrolled coronary disease or New York Heart Association (NYHA) class III-IV heart disease.
* Known infection with human immunodeficiency virus (HIV), hepatitis B or C.
* Pregnant or lactating women.
* Presence of active 2nd malignancy requiring treatment. 2nd malignancies with low activity which do not require treatment (i.e., low grade prostate cancer, basal cell or squamous cell skin cancer) do not constitute exclusions.
* Inability to comply with study and/or follow-up procedures.
* Presence of central nervous system (CNS) disease
* Patients with history of non-response to both pentostatin plus rituximab and to bendamustine plus rituximab.
* Receipt of a live vaccine within 4 weeks prior to randomization. Efficacy and/or safety of immunization during periods of B-cell depletion have not been adequately studied. It is recommended that a patients vaccination record and possible requirements be reviewed. The patient may have any required vaccination/booster administered at least 4 weeks prior to the initiation of study treatment. Review of the patient's immunization status for the following vaccinations is recommended: tetanus; diphtheria; influenza; Pneumococcal polysaccharide; Varicella; measles, mumps and rubella (MMR); and hepatitis B. Patients who are considered to be at high risk for hepatitis B virus (HBV) infection and for whom the investigator has determined that immunization is indicated should complete the entire HBV vaccine series at least 4 weeks prior to participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2010-07-01 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2027-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Kreitman, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI).

REFERENCES:
- [Background] Bouroncle BA. Thirty-five years in the progress of hairy cell leukemia. Leuk Lymphoma. 1994;14 Suppl 1:1-12. PMID 7820038
- [Background] Kreitman RJ, Cheson BD. Malignancy: Current Clinical Practice: Treatment of Hairy Cell Leukemia at the Close of the 20th Century. Hematology. 1999;4(4):283-303. doi: 10.1080/10245332.1999.11746452. PMID 11399570
- [Background] Jemal A, Siegel R, Ward E, Murray T, Xu J, Thun MJ. Cancer statistics, 2007. CA Cancer J Clin. 2007 Jan-Feb;57(1):43-66. doi: 10.3322/canjclin.57.1.43. PMID 17237035
- [Derived] Schroeder B, Yuan CM, Wang HW, Mohindroo C, Zhou H, Raffeld M, Xi L, Arons E, Feurtado JC, James-Echenique L, Calvo KR, Maric I, Kreitman RJ. Phase 2 trial of rituximab with either pentostatin or bendamustine for multiply relapsed or refractory hairy cell leukemia. Blood. 2025 Oct 8:blood.2025031243. doi: 10.1182/blood.2025031243. Online ahead of print. PMID 41060318
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2010-C-0025.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-Randomized to 70 mg/m2 Bendamustine-Rituximab: Treatment Assignment Code 5 (TAC 5) Rituximab + Bendamustine at 70 mg/m^2 for initial tolerability study (closed) Rituximab 375 mg/m^2 on day 1, 15 for 6 x 28-day cycles 6 participants to bendamustine 70 mg/m^2/day, days 1 and 2 each cycle Acetaminophen: Treatment of infusion-related symptoms with acetaminophen is recommended.
  Diphenhydramine: Treatment of infusion-related symptoms with diphenhydramine is recommended.
  Epinephrine: Epinephrine should be available for immediate use in the event of a hypersensitivity reaction to Rituximab.
  Antihistamines: Antihistamines should be available for immediate use in the event of a hypersensitivity reaction to Rituximab.
  Corticosteroids: Corticosteroids should be available for immediate use in the event of a hypersensitivity reaction to Rituximab.
  Bronchodilators: Additional treatment with bronchodilators may be indicated. Intravenous (IV) Saline: Additional treatment with intravenous (IV) saline may be indicated.
- Non-randomized to 90 mg/m^2 Bendamustine-Rituximab: Treatment Assignment Code 5 (TAC 5) Rituximab + Bendamustine at 90 mg/m^2 for initial tolerability study (closed) Rituximab 375 mg/m^2 on day 1, 15 for 6 x 28-day cycles Bendamustine: 6 participants to bendamustine 90 mg/m^2/day, days 1 and 2 each cycle Acetaminophen: Treatment of infusion-related symptoms with acetaminophen is recommended.
  Diphenhydramine: Treatment of infusion-related symptoms with diphenhydramine is recommended.
  Epinephrine: Epinephrine should be available for immediate use in the event of a hypersensitivity reaction to Rituximab.
  Antihistamines: Antihistamines should be available for immediate use in the event of a hypersensitivity reaction to Rituximab.
  Corticosteroids: Corticosteroids should be available for immediate use in the event of a hypersensitivity reaction to Rituximab.
  Bronchodilators: Additional treatment with bronchodilators may be indicated. Intravenous (IV) Saline: Additional treatment with intravenous (IV) saline may be indicated
- Randomized to 90 mg/m^2 Bendamustine-Rituximab: Treatment Assignment Code 5 (TAC 5) Rituximab + Bendamustine at 90 mg/m^2 Rituximab: 28 participants Rituximab 375 mg/m^2 on day 1, 15 for 6 x 28-day cycles Bendamustine:28 participants to bendamustine 90 mg/m^2/day, days 1 and 2 each cycle, days 1 and 2 each cycle Acetaminophen: Treatment of infusion-related symptoms with acetaminophen is recommended.
  Diphenhydramine: Treatment of infusion-related symptoms with diphenhydramine is recommended.
  Epinephrine: Epinephrine should be available for immediate use in the event of a hypersensitivity reaction to Rituximab.
  Antihistamines: Antihistamines should be available for immediate use in the event of a hypersensitivity reaction to Rituximab.
  Corticosteroids: Corticosteroids should be available for immediate use in the event of a hypersensitivity reaction to Rituximab.
  Bronchodilators: Additional treatment with bronchodilators may be indicated. Intravenous (IV) Saline: Additional treatment with intravenous (IV) saline may be indicated.
- Randomized to Pentostatin-Rituximab: Treatment Assignment Code 2 (TAC 2) Rituximab + Pentostatin
  Pentostatin: 28 participants to pentostatin 4 mg/m^2 days 1 and 15 of each cycle.
  Rituximab: Rituximab 375 mg/m^2 on day 1, 15 for 6 x 28-day cycles
  Acetaminophen: Treatment of infusion-related symptoms with acetaminophen is recommended.
  Diphenhydramine: Treatment of infusion-related symptoms with diphenhydramine is recommended.
  Epinephrine: Epinephrine should be available for immediate use in the event of a hypersensitivity reaction to Rituximab.
  Antihistamines: Antihistamines should be available for immediate use in the event of a hypersensitivity reaction to Rituximab.
  Corticosteroids: Corticosteroids should be available for immediate use in the event of a hypersensitivity reaction to Rituximab.
  Bronchodilators: Additional treatment with bronchodilators may be indicated.
  Intravenous (IV) Saline: Additional treatment with intravenous (IV) saline may be indicated.
- Non-randomized to Bendamustine 90mg/m^2 or Pentostatin 4mg/m^2 With Rituximab: Treatment Assignment Code 5 (TAC 5) Rituximab + Bendamustine at 90 mg/m^2 or Rituxan + Pentostatin After initial tolerability studies are completed. Non-randomize up to 4 total participants to Bendamustine and/or Pentostatin with Rituximab Rituximab 375 mg/m^2 on day 1, 15 for 6 x 28-day cycles Bendamustine: 1-4 participants to bendamustine 90 mg/m^2/day, days 1 and 2 each cycle Pentostatin 1-4 participants to pentostatin 4 mg/m^2 days 1 and 15 of each cycle.
  Acetaminophen: Treatment of infusion-related symptoms with acetaminophen is recommended.
  Diphenhydramine: Treatment of infusion-related symptoms with diphenhydramine is recommended.
  Epinephrine: Epinephrine should be available for immediate use in the event of a hypersensitivity reaction to Rituximab.
  Antihistamines: Antihistamines should be available for immediate use in the event of a hypersensitivity reaction to Rituximab.
  Corticosteroids: Corticosteroids should be available for immediate use in the event of a hypersensitivity reaction to Rituximab.
  Bronchodilators: Additional treatment with bronchodilators may be indicated. Intravenous (IV) Saline: Additional treatment with intravenous (IV) saline may be indicated.
Period: Overall Study
Arm/Group | Non-Randomized to 70 mg/m2 Bendamustine-Rituximab | Non-randomized to 90 mg/m^2 Bendamustine-Rituximab | Randomized to 90 mg/m^2 Bendamustine-Rituximab | Randomized to Pentostatin-Rituximab | Non-randomized to Bendamustine 90mg/m^2 or Pentostatin 4mg/m^2 With Rituximab
Started | 6 | 6 | 28 | 28 | 1
Completed | 6 | 6 | 24 | 27 | 1
Not Completed | 0 | 0 | 4 | 1 | 0
Not completed — Did not receive 6 cycles. | 0 | 0 | 4 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-Randomized to 70 mg/m2 Bendamustine-Rituximab | Non-randomized to 90 mg/m^2 Bendamustine-Rituximab | Randomized to 90 mg/m^2 Bendamustine-Rituximab | Randomized to Pentostatin-Rituximab | Non-randomized to Bendamustine 90mg/m^2 or Pentostatin 4mg/m^2 With Rituximab | Total
Number analyzed (Participants) | 6 | 6 | 28 | 28 | 1 | 69
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 6 | 16 | 15 | 0 | 39
  >=65 years | 4 | 0 | 12 | 13 | 1 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.65 (3.03) | 58.67 (3.14) | 61.87 (9.75) | 61.55 (12.23) | 71.2 (0) | 62.01 (10.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 6 | 4 | 0 | 12
  Male | 4 | 6 | 22 | 24 | 1 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 28 | 26 | 1 | 67
  Unknown or Not Reported | 0 | 0 | 0 | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 1 | 0 | 3
  White | 6 | 5 | 26 | 27 | 1 | 65
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 28 | 28 | 1 | 69

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Receiving Pentostatin + Rituximab and Bendamustine + Rituximab Who Achieve a Complete Remission (CR) + Partial Response (PR)
Description: Number of participants receiving pentostatin + rituximab and bendamustine + rituximab who achieve a CR +PR measured by the following response criteria. Complete remission is all of the following for at least 4 weeks: absolute neutrophil count ≥ 1500/mm^3, platelets ≥ 100,000/mm^3, hemoglobin ≥ 11g/dl, spleen non-palpable below the costal margin, or not below costal margin on computed tomography, and circulating hairy cell leukemia (HCL) cells either non-visible on Wright stain or < 1% by flow cytometry. Partial response is all of the following for at least 4 weeks: neutrophils ≥ 1,500/µL or 50% improvement over baseline, platelets ≥100,000/µL or 50% improvement over baseline, hemoglobin ≥ 11.0 g/dL or 50% improvement over baseline, ≥ 50% decrease in circulating malignant HCL count from the pretreatment baseline, ≥ 50% reduction in sum of products of perpendicular diameters or decrease to ≤ 2 cm in evaluable (> 2cm) lymphadenopathy.
Time Frame: At end of treatment, approximately 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Non-Randomized to 70 mg/m2 Bendamustine-Rituximab | Non-randomized to 90 mg/m^2 Bendamustine-Rituximab | Randomized to 90 mg/m^2 Bendamustine-Rituximab | Randomized to Pentostatin-Rituximab | Non-randomized to Bendamustine 90mg/m^2 or Pentostatin 4mg/m^2 With Rituximab
Number analyzed (Participants) | 6 | 6 | 28 | 28 | 1
Participants
  Complete Remission | 3 | 4 | 20 | 22 | 1
  Partial Response | 3 | 2 | 4 | 4 | 0

2. Secondary Outcome: Pentostatin + Rituximab and Bendamustine + Rituximab in Crossover When Used After Failure of the 1st Regimen
Description: Compare the 2 regimens - pentostatin + rituximab and bendamustine + rituximab in crossover when used after failure of the 1st regimen.
Time Frame: 4 years
Reporting Status: Not Posted, anticipated posting 2027-12

3. Secondary Outcome: Response Rate
Description: Response rate between participants who received rituximab plus either pentostatin or bendamustine measured by the following response criteria. Complete remission is all of the following for at least 4 weeks: absolute neutrophil count ≥ 1500/mm^3, platelets ≥ 100,000/mm^3, hemoglobin ≥ 11g/dl, spleen non-palpable below the costal margin, or not below costal margin on computed tomography, and circulating hairy cell leukemia (HCL) cells either non-visible on Wright stain or < 1% by flow cytometry. Partial response is all of the following for at least 4 weeks: neutrophils ≥ 1,500/µL or 50% improvement over baseline, platelets ≥100,000/µL or 50% improvement over baseline, hemoglobin ≥ 11.0 g/dL or 50% improvement over baseline, ≥ 50% decrease in circulating malignant HCL count from the pretreatment baseline, ≥ 50% reduction in sum of products of perpendicular diameters. Progressive disease is appearance of new evaluable lymph nodes >2cm. Stable disease is none of the above
Time Frame: 4 years
Reporting Status: Not Posted, anticipated posting 2027-11

4. Secondary Outcome: Mechanism of Thrombocytopenia
Description: The mechanism of thrombocytopenia after purine analog plus rituximab.
Time Frame: 4 years
Reporting Status: Not Posted, anticipated posting 2027-12

5. Secondary Outcome: Hairy Cell Leukemia (HCL) Biology
Description: HCL biology was determined by cloning, sequencing and characterizing monoclonal immunoglobulin rearrangements, and other genes.
Time Frame: 4 years
Reporting Status: Not Posted, anticipated posting 2027-12

6. Secondary Outcome: Correlation of Measurable Residual Disease (MRD) Levels and Tumor Markers With Response
Description: Determine if MRD levels and tumor markers (soluble cluster of Differentiation 25 (CD25) and cluster of differentiation-22 (CD22), and real-time quantitative reverse transcriptase polymerase chain reaction (RQ-PCR) correlate with response and clinical endpoints, and if bone marrow magnetic resonance imaging (MRI) signal correlates with bone marrow biopsy (BMBx) results, and whether these tests could in some cases possibly replace BMBx.
Time Frame: 4 years
Reporting Status: Not Posted, anticipated posting 2027-12

7. Secondary Outcome: Measurable Residual Disease (MRD)-Free Survival
Description: MRD-free survival is defined by the Response criteria.
Time Frame: 4 years
Reporting Status: Not Posted, anticipated posting 2027-12

8. Secondary Outcome: Disease-free Survival (DFS)
Description: Disease-free survival is the time from start of treatment to documented evidence of disease progression measured by the following response criteria. Progressive disease ≥50% increase in sum of products of perpendicular diameters of evaluable (> 2cm) lymphadenopathy or appearance of new evaluable lymph nodes >2cm.
Time Frame: time from start of treatment to documented evidence of disease progression
Reporting Status: Not Posted, anticipated posting 2027-12

9. Secondary Outcome: Overall Survival
Description: OS is the time between the first day of treatment to the day of death.
Time Frame: time between the first day of treatment to the day of death
Reporting Status: Not Posted, anticipated posting 2027-12

10. Secondary Outcome: Toxicity
Description: Toxicity was assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: 4 years
Reporting Status: Not Posted, anticipated posting 2027-12

11. Secondary Outcome: Cluster of Differentiation 4 (CD4+) T-cells
Description: Cluster of differentiation 4 (CD4+) T-cells assessed by analysis.
Time Frame: 4 years
Reporting Status: Not Posted, anticipated posting 2027-12

12. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 103 months and 19 days; 133 months and 11 days; 111 months and 15 days; 102 months and 25 days; 44 months and 14 days; and 19 months and 2 days for each group respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Non-Randomized to 70 mg/m2 Bendamustine-Rituximab | Non-randomized to 90 mg/m^2 Bendamustine-Rituximab | Randomized to 90 mg/m^2 Bendamustine-Rituximab | Randomized to Pentostatin-Rituximab | Non-randomized to Bendamustine 90mg/m^2 or Pentostatin 4mg/m^2 With Rituximab
Number analyzed (Participants) | 6 | 6 | 28 | 28 | 1
Participants | 6 | 6 | 28 | 28 | 1

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 103 months and 19 days; 133 months and 11 days; 111 months and 15 days; 102 months and 25 days; 44 months and 14 days; and 19 months and 2 days for each group respectively.
Arm/Group | Non-Randomized to 70 mg/m2 Bendamustine-Rituximab | Non-randomized to 90 mg/m^2 Bendamustine-Rituximab | Randomized to 90 mg/m^2 Bendamustine-Rituximab | Randomized to Pentostatin-Rituximab | Non-randomized to Bendamustine 90mg/m^2 or Pentostatin 4mg/m^2 With Rituximab
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 3/28 | 5/28 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 8/28 | 7/28 | 0/1
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 28/28 | 28/28 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-Randomized to 70 mg/m2 Bendamustine-Rituximab (N=6) | Non-randomized to 90 mg/m^2 Bendamustine-Rituximab (N=6) | Randomized to 90 mg/m^2 Bendamustine-Rituximab (N=28) | Randomized to Pentostatin-Rituximab (N=28) | Non-randomized to Bendamustine 90mg/m^2 or Pentostatin 4mg/m^2 With Rituximab (N=1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Allergic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Edema face (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (3) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Vasovagal reaction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-Randomized to 70 mg/m2 Bendamustine-Rituximab (N=6) | Non-randomized to 90 mg/m^2 Bendamustine-Rituximab (N=6) | Randomized to 90 mg/m^2 Bendamustine-Rituximab (N=28) | Randomized to Pentostatin-Rituximab (N=28) | Non-randomized to Bendamustine 90mg/m^2 or Pentostatin 4mg/m^2 With Rituximab (N=1)
Abdominal pain (Gastrointestinal disorders) | 5 (10) | 2 (2) | 5 (5) | 5 (7) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 5 (15) | 2 (3) | 13 (23) | 11 (18) | 0 (0)
Alkaline phosphatase increased (Investigations) | 3 (8) | 2 (5) | 8 (15) | 5 (7) | 1 (1)
Allergic reaction (Immune system disorders) | 4 (8) | 0 (0) | 8 (9) | 3 (6) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 4 (9) | 10 (26) | 6 (12) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 7 (13) | 4 (5) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (4) | 1 (1) | 2 (4) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (4) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 5 (18) | 3 (4) | 18 (27) | 9 (16) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 6 (8) | 7 (9) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 3 (10) | 1 (1) | 6 (14) | 5 (14) | 0 (0)
Blurred vision (Eye disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (2) | 2 (5) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
CD4 lymphocytes decreased (Investigations) | 1 (1) | 0 (0) | 4 (9) | 6 (17) | 0 (0)
CPK increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Carbon monoxide diffusing capacity decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac disorders - Other, QTC Interval prolonged (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 2 (3) | 2 (3) | 0 (0)
Chills (General disorders) | 5 (9) | 4 (9) | 13 (30) | 19 (35) | 0 (0)
Cholesterol high (Investigations) | 0 (0) | 0 (0) | 2 (2) | 3 (5) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (1) | 8 (9) | 9 (18) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 14 (19) | 13 (15) | 0 (0)
Creatinine increased (Investigations) | 1 (2) | 2 (2) | 7 (14) | 3 (7) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (6) | 1 (1) | 7 (11) | 11 (17) | 0 (0)
Dizziness (Nervous system disorders) | 1 (2) | 1 (1) | 6 (8) | 5 (5) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Dysgeusia (Nervous system disorders) | 3 (8) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (3) | 3 (6) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1) | 9 (14) | 8 (15) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Edema face (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 2 (3) | 3 (3) | 4 (4) | 7 (7) | 0 (0)
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Eye disorders - Other, Hemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (3) | 0 (0)
Facial pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (2) | 10 (11) | 7 (14) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (4) | 7 (12) | 8 (10) | 0 (0)
Fever (General disorders) | 2 (3) | 3 (3) | 15 (26) | 11 (19) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Floaters (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flu like symptoms (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 1 (2) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
GGT increased (Investigations) | 1 (1) | 1 (2) | 4 (4) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haptoglobin decreased (Investigations) | 0 (0) | 0 (0) | 5 (7) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 2 (3) | 3 (3) | 15 (27) | 9 (25) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Hemoglobin increased (Investigations) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Hemoglobinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (7) | 3 (5) | 14 (30) | 9 (20) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1) | 4 (7) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 1 (1) | 3 (5) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 4 (6) | 3 (3) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 5 (5) | 1 (1) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (7) | 3 (4) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 4 (5) | 4 (7) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (15) | 2 (8) | 10 (29) | 13 (35) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 4 (6) | 5 (5) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (2) | 3 (3) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 4 (9) | 4 (9) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 1 (3) | 7 (11) | 5 (8) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 2 (3) | 3 (4) | 5 (7) | 10 (16) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 7 (9) | 6 (8) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 1 (1) | 5 (5) | 6 (6) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, Upper Respiratory (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (General disorders) | 1 (2) | 1 (1) | 1 (2) | 6 (24) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (3) | 2 (2) | 0 (0)
Investigations - Other, Creatinine decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Irregular menstruation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 23 (135) | 22 (132) | 0 (0)
Lymphocyte count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metabolism and nutrition disorders - Other, Bicarbonate increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (4) | 6 (17) | 10 (13) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (5) | 2 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (16) | 3 (8) | 21 (44) | 19 (53) | 0 (0)
Neck edema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (5) | 3 (14) | 15 (35) | 15 (61) | 0 (0)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 9 (11) | 3 (3) | 0 (0)
Oral pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Pain (General disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 8 (8) | 4 (5) | 0 (0)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Papulopustular rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 1 (1) | 3 (3) | 4 (5) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Platelet count decreased (Investigations) | 4 (17) | 5 (9) | 19 (57) | 14 (32) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3) | 3 (3) | 6 (9) | 7 (13) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 2 (2) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (3) | 3 (5) | 6 (9) | 10 (22) | 0 (0)
Scrotal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Serum amylase increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 2 (3) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (4) | 3 (3) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Superficial thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 2 (2) | 5 (6) | 3 (3) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Uveitis (Eye disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal inflammation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (5) | 1 (1) | 10 (21) | 10 (19) | 0 (0)
Watering eyes (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Weight gain (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight loss (Investigations) | 1 (1) | 1 (1) | 3 (4) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 4 (13) | 4 (16) | 15 (118) | 21 (90) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye disorders - Other, Macular degeneration (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Investigations - Other, Increased prothrombin time (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2022-09-06): https://cdn.clinicaltrials.gov/large-docs/86/NCT01059786/Prot_SAP_000.pdf
  • Informed Consent Form: Cohort Eligibility Consent (2022-10-11): https://cdn.clinicaltrials.gov/large-docs/86/NCT01059786/ICF_001.pdf
  • Informed Consent Form: Affected Patients Consent (2022-10-11): https://cdn.clinicaltrials.gov/large-docs/86/NCT01059786/ICF_002.pdf